CLINICAL TRIAL: NCT02951988
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter Study of Rapastinel as Adjunctive Therapy in the Prevention of Relapse in Patients With Major Depressive Disorder
Brief Title: A Study of Rapastinel as Adjunctive Therapy in the Prevention of Relapse in Patients With Major Depressive Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Naurex, Inc, an affiliate of Allergan plc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RAP-MD-04
Record Dates: First submitted 2016-10-31; First posted 2016-11-01 (Estimated); Results first posted 2020-03-09 (Actual); Last update posted 2020-03-09 (Actual); Status verified 2020-02

CONDITIONS: Depressive Disorder, Major
MeSH Terms: conditions — Depressive Disorder, Major | interventions — GLYX-13 peptide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Rapastinel 450 mg Weekly (Experimental): Rapastinel 450 milligrams (mg) intravenous (IV) once a week during OLTP followed by rapastinel 450 mg IV once a week during DBTP.
  Interventions: Drug: Rapastinel
- Rapastinel 450 mg Every 2 Weeks (Experimental): Rapastinel 450 mg IV once a week during OLTP followed by rapastinel 450 mg IV once every 2 weeks during DBTP.
  Interventions: Drug: Rapastinel
- Placebo (Placebo Comparator): Rapastinel 450 mg IV once a week during OLTP followed by placebo-matching rapastinel 450 mg IV once a week during DBTP.
  Interventions: Drug: Placebo-matching Rapastinel

INTERVENTIONS:
Drug: Rapastinel — Rapastinel pre-filled syringes for IV injections.
  Arms: Rapastinel 450 mg Every 2 Weeks; Rapastinel 450 mg Weekly
Drug: Placebo-matching Rapastinel — Placebo-matching rapastinel pre-filled syringes for weekly IV injections.
  Arms: Placebo

SUMMARY:
This study will evaluate the efficacy, safety and tolerability of rapastinel 450 milligrams (mg) intravenous (IV) once weekly or once every 2 weeks versus placebo as an adjunctive treatment to ongoing anti-depressive therapy (ADT) in the prevention of relapse in participants with Major Depressive Disorder (MDD).

ELIGIBILITY:
Inclusion Criteria:

* Meet Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria for MDD
* Current major depressive episode of at least 8 weeks and not exceeding 18 months in duration at Screening
* Have no more than partial response (< 50% improvement) to ongoing treatment with a protocol-allowed antidepressant
* If female of childbearing potential, have a negative serum β-human chorionic gonadotropin (β-hCG) pregnancy test.

Exclusion Criteria:

* DSM-5-based diagnosis of any disorder other than MDD that was the primary focus of treatment within 6 months before Screening
* Lifetime history of meeting DSM-5 criteria for:
* Schizophrenia spectrum or other psychotic disorder
* Bipolar or related disorder
* Major neurocognitive disorder
* Neurodevelopmental disorder of greater than mild severity or of a severity that impacts the participant's ability to consent, follow study directions, or otherwise safely participate in the study
* Dissociative disorder
* Posttraumatic stress disorder
* MDD with psychotic features
* Significant suicide risk, as judged by the Investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1304 (Actual)
Dates: Start 2016-11-13 (Actual); Primary Completion 2019-02-22 (Actual); Study Completion 2019-02-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jenna Hoogerheyde, Study Director — Allergan
Locations (137):
- United States (137):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Harmonex Neuroscience Research, Dothan, Alabama
  - NoesisPharma, Phoenix, Arizona
  - University of Arizona Department of Psychiatry, Tucson, Arizona
  - Woodland International Research Group, Little Rock, Arkansas
  - Woodland Research Northwest, Rogers, Arkansas
  - California Pharmaceutical Research Institute, Inc, Anaheim, California
  - Southern California Research LLC., Beverly Hills, California
  - ATP Clinical Research Inc., Costa Mesa, California
  - ProScience Research Group, Culver City, California
  - Pharmacology Research Institute, Encino, California
  - Collaborative Neuroscience Network, LLC, Garden Grove, California
  - Behavioral Research Specialists, LLC, Glendale, California
  - Sun Valley Research Center, Imperial, California
  - Irvine Center for Clinical Research, Inc, Irvine, California
  - Synergy Clinical Research Center of Escondido, Lemon Grove, California
  - Synergy San Diego, Lemon Grove, California
  - Pharmacology Research Institute, Los Alamitos, California
  - Pacific Research Partners; LLC., Oakland, California
  - Excell Research, Oceanside, California
  - NRC Research Institute, Orange, California
  - Asclepes Research Centers, Panorama City, California
  - Anderson Clinical Research, Redlands, California
  - CITrials, Riverside, California
  - Artemis Institute for Clinical Research, San Diego, California
  - PCSD Feighner Research, San Diego, California
  - Artemis Institute for Clinical Research, San Marcos, California
  - Thomas M. Shiovitz, M.D., Inc., DBA California Neuroscience Research Medical Group, Inc.,, Sherman Oaks, California
  - Viking Clinical Research, Temecula, California
  - Pacific Clinical Research Medical, Upland, California
  - MCB Clinical Research Center, Colorado Springs, Colorado
  - Comprehensive Psychiatric Care, Norwich, Connecticut
  - Meridien Research, Bradenton, Florida
  - Gulfcoast Clinical Research Center, Fort Myers, Florida
  - Sarkis Clinical Trials, Gainesville, Florida
  - MD Clinical, Hallandale, Florida
  - Reliable Clinical Research, Hialeah, Florida
  - Advanced Research Institute of Miami, Homestead, Florida
  - Clinical Neuroscience Solutions, Inc, Jacksonville, Florida
  - Meridien Research, Lakeland, Florida
  - Innovative Clinical Research, Inc, Lauderhill, Florida
  - Innova Clinical Trials Inc., Miami, Florida
  - International Research Associates, LLC, Miami, Florida
  - Research Centers of America, Oakland Park, Florida
  - Sarkis Clinical Trials, Ocala, Florida
  - Medical Research Group of Central Florida, Orange City, Florida
  - Clinical Neuroscience Solutions, Inc, Orlando, Florida
  - Combined Research Orlando Phase I-IV, Orlando, Florida
  - Millenia Psychiatry & Research, Inc, Orlando, Florida
  - Olympian Clinical Research, Tampa, Florida
  - The University of South Florida Board of Trustees, A public Body Corporate, for University of South Florida, Tampa, Florida
  - Institute for Advanced Medical Research, Alpharetta, Georgia
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - iResearch Atlanta, LLC, Decatur, Georgia
  - Northwest Behavioral Research Center, Marietta, Georgia
  - IRIS Research, Smyrna, Georgia
  - Great Lakes Clinical Trials, Chicago, Illinois
  - Alexian Brothers Center for Psychiatric Research, Hoffman Estates, Illinois
  - Capstone Clinical Research, Libertyville, Illinois
  - AMR - Baber Research, Inc., Naperville, Illinois
  - Psychiatric Associates, Overland Park, Kansas
  - Phoenix Medical Research, Prairie Village, Kansas
  - Heartland Research Associates, Wichita, Kansas
  - Lake Charles Clinical Trials, Lake Charles, Louisiana
  - Louisiana Clinical Research, Shreveport, Louisiana
  - J Gary Booker, MD APMC, Shreveport, Louisiana
  - Sheppard Pratt Health System, Baltimore, Maryland
  - Pharmasite Research, Inc, Baltimore, Maryland
  - CBH Health, Rockville, Maryland
  - Boston Clinical Trials, Boston, Massachusetts
  - ActivMed Practices & Research, Inc., Methuen, Massachusetts
  - BTC of New Bedford, New Bedford, Massachusetts
  - Adams Clinical Trials, Watertown, Massachusetts
  - Coastal Research Associates, Weymouth, Massachusetts
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - Precise Research Centers, Flowood, Mississippi
  - Millennium Psychiatric Associates, Creve Coeur, Missouri
  - Psychiatric Care and Research Center, O'Fallon, Missouri
  - St. Charles Psychiatric Associates - Midwest Research Group, Saint Charles, Missouri
  - Alivation Research, Lincoln, Nebraska
  - Altea Research, Las Vegas, Nevada
  - Healthy Perspectives - Innovative Mental Health Services. PLLC, Nashua, New Hampshire
  - Hassman Research Institute, LLC, Berlin, New Jersey
  - Center for Emotional Fitness, Cherry Hill, New Jersey
  - Pharmaceutical Research Associates Inc, Marlton, New Jersey
  - Global Medical Institute, LLC, Princeton, New Jersey
  - Bio Behavioral Health, Toms River, New Jersey
  - Albuquerque Neuroscience, Inc, Albuquerque, New Mexico
  - SPRI Clinical Trials, Inc, Brooklyn, New York
  - Bioscience Research, Mount Kisco, New York
  - Manhattan Behavioral Medicine, New York, New York
  - Eastside Comprehensive Medical Center, LLC, New York, New York
  - The Medical Research Network, LLC, New York, New York
  - Fieve Clinical Research, New York, New York
  - Finger Lakes Clinical Research, Rochester, New York
  - Richmond Behavioral Associates, Staten Island, New York
  - New Hope Clinical Research Inc., Charlotte, North Carolina
  - Richard H. Weisler, MD, PA, Raleigh, North Carolina
  - Neuro-Behavioral Clinical Research, Inc, Canton, Ohio
  - Patient Priority Clinical Site, LLC, Cincinnati, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - The Ohio State University Department of Psychiatry, Columbus, Ohio
  - Midwest Clinical Research Center LLC, Dayton, Ohio
  - Charak Clinical Research Center, Garfield Heights, Ohio
  - Lindner Center of Hope, Mason, Ohio
  - Professional Psychiatric Services, Mason, Ohio
  - IPS Research, Oklahoma City, Oklahoma
  - Red River Medical Research Center, LLC, Oklahoma City, Oklahoma
  - Sooner Clinical Research, Inc, Oklahoma City, Oklahoma
  - Paradigm Research Professionals, Oklahoma City, Oklahoma
  - Summit Research Network, Portland, Oregon
  - Lehigh Center for Clinical Research, Allentown, Pennsylvania
  - Suburban Research Associates, Media, Pennsylvania
  - Dr. Cherian Verghese, Norristown, Pennsylvania
  - Carolina Clinical Trials, Inc., Charleston, South Carolina
  - Coastal Carolina Research Center, Inc., Mt. Pleasant, South Carolina
  - Clinical Neuroscience Solutions, Inc, Memphis, Tennessee
  - Research Strategies of Memphis, LLC, Memphis, Tennessee
  - Donald J. Garcia, Jr., MD, PA, Austin, Texas
  - Community Clinical Research, Inc., Austin, Texas
  - BioBehavioral Research of Austin, Austin, Texas
  - Houston Clinical Trials, LLC, Bellaire, Texas
  - Relaro Medical Trials, Dallas, Texas
  - El Campo Clinical Trials, El Campo, Texas
  - North Texas Clinical Trials, Fort Worth, Texas
  - Earle Research, Houston, Texas
  - Red Oak Psychiatry Associates, PA, Houston, Texas
  - Clinical Trials of Texas, San Antonio, Texas
  - Family Psychiatry of The Wood, The Woodlands, Texas
  - Grayline Clinical Drug Trials, Wichita Falls, Texas
  - Psychiatric and Behavioral Solutions, Salt Lake City, Utah
  - PRA Health Sciences, Salt Lake City, Utah
  - Department of Psychiatry and Neurobehavioral Sciences, University of Virginia, Charlottesville, Virginia
  - Psychiatric Alliance of the Blue Ridge, Inc, Charlottesville, Virginia
  - NorthWest Clinical Research Center, Bellevue, Washington
  - Pacific Institute of Medical Sciences, Bothell, Washington
  - Eastside Therapeutic Resource, Everett, Washington

REFERENCES:
- See also: More Information — http://www.allerganclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients from RAP-MD-04, completed 1 of the rapastinel lead-in studies - RAP-MD-01, RAP-MD-02, or RAP-MD-03.
Pre-assignment Details: A total of 1304 patients enrolled in the Open Label Treatment Period (OLTP). Of these, 1056 completed the OLTP and 604 entered the Double Blind Treatment Period (DBTP) and were randomized.
Groups:
- OLTP Rapastinel 450 mg Weekly + ADT: Rapastinel 450 milligrams (mg) intravenous (IV) once a week during OLTP.
- DBTP Placebo: Rapastinel 450 mg IV once a week during OLTP followed by placebo-matching rapastinel 450 mg IV once a week during DBTP.
- DBTP Rapastinel 450 mg Every 2 Weeks: Rapastinel 450 mg IV once a week during OLTP followed by rapastinel 450 mg IV once every 2 weeks.
- DBTP Rapastinel 450 mg Weekly: Rapastinel 450 mg IV once a week during OLTP followed by rapastinel 450 mg IV once a week during DBTP.
Period: Open-Label Treatment Period
Arm/Group | OLTP Rapastinel 450 mg Weekly + ADT | DBTP Placebo | DBTP Rapastinel 450 mg Every 2 Weeks | DBTP Rapastinel 450 mg Weekly
Started | 1304 | 0 | 0 | 0
Completed | 1056 | 0 | 0 | 0
Not Completed | 248 | 0 | 0 | 0
Not completed — Miscellaneous Reasons | 8 | 0 | 0 | 0
Not completed — Study terminated by sponsor | 9 | 0 | 0 | 0
Not completed — Non-compliance with background ADT | 2 | 0 | 0 | 0
Not completed — Non-compliance with study drug | 5 | 0 | 0 | 0
Not completed — Protocol Violation | 22 | 0 | 0 | 0
Not completed — Pregnancy | 2 | 0 | 0 | 0
Not completed — Lost to Follow-up | 28 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 78 | 0 | 0 | 0
Not completed — Lack of Efficacy | 49 | 0 | 0 | 0
Not completed — Adverse Event | 45 | 0 | 0 | 0
Period: Double-Blind Treatment Period
Arm/Group | OLTP Rapastinel 450 mg Weekly + ADT | DBTP Placebo | DBTP Rapastinel 450 mg Every 2 Weeks | DBTP Rapastinel 450 mg Weekly
Started | 0 | 202 | 202 | 200
Completed | 0 | 101 | 101 | 85
Not Completed | 0 | 101 | 101 | 115
Not completed — Site terminated by sponsor | 0 | 0 | 1 | 1
Not completed — Study terminated by sponsor | 0 | 58 | 54 | 69
Not completed — Non-compliance with study drug | 0 | 1 | 3 | 0
Not completed — Protocol Violation | 0 | 4 | 4 | 8
Not completed — Pregnancy | 0 | 1 | 1 | 0
Not completed — Lost to Follow-up | 0 | 4 | 12 | 3
Not completed — Withdrawal by Subject | 0 | 23 | 22 | 28
Not completed — Adverse Event | 0 | 8 | 3 | 6
Not completed — Miscellaneous Reasons | 0 | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Double-blind modified Intent-to-Treat Population consists of all patients in the Open-label Safety Population who were randomized to a treatment group during the DBTP of the study and received at least 1 dose of IP during the DBTP.
Groups:
- Rapastinel 450 mg Weekly: Rapastinel 450 mg IV once a week during OLTP followed by rapastinel 450 mg IV once a week during DBTP.
- Total: Total of all reporting groups
Arm/Group | Placebo | Rapastinel 450 mg Every 2 Weeks | Rapastinel 450 mg Weekly | Total
Number analyzed (Participants) | 202 | 202 | 200 | 604
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.2 (12.45) | 45.4 (12.17) | 44.7 (12.15) | 45.1 (12.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 148 | 142 | 152 | 442
  Male | 54 | 60 | 48 | 162
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 25 | 29 | 29 | 83
  Not Hispanic or Latino | 177 | 173 | 171 | 521
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 162 | 170 | 162 | 494
  Black or African American | 35 | 27 | 29 | 91
  Asian | 4 | 4 | 2 | 10
  American Indian or Alaska Native | 0 | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 3 | 3
  Multiple | 1 | 1 | 2 | 4
Weight [Mean (Standard Deviation); unit: kg] | 86.49 (19.15) | 88.29 (18.78) | 85.39 (17.46) | 86.73 (18.49)
Height [Mean (Standard Deviation); unit: cm] | 167.27 (8.85) | 168.12 (9.78) | 167.36 (9.13) | 167.58 (9.25)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 30.94 (6.74) | 31.33 (6.83) | 30.45 (5.69) | 30.91 (6.44)

OUTCOME MEASURES:

1. Primary Outcome: Time to First Relapse During the First 52 Weeks of the Double-Blind Treatment Period
Description: The time in days to first relapse is defined as the number of days from the date of randomization to the first relapse.
Time Frame: 52 Weeks
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Placebo | Rapastinel 450 mg Every 2 Weeks | Rapastinel 450 mg Weekly
Number analyzed (Participants) | 202 | 202 | 200
Days | 232 [167 to NA] — Not enough events to allow the estimation of the percentiles and the standard error for the confidence intervals. | 225 [127 to 323] | 336 [157 to NA] — Not enough events to allow the estimation of the percentiles and the standard error for the confidence intervals.
Statistical Analysis 1: Comparison: Placebo vs Rapastinel 450 mg Every 2 Weeks; Test type: Superiority; p = 0.5305, Log Rank
Statistical Analysis 2: Comparison: Placebo vs Rapastinel 450 mg Weekly; Test type: Superiority; p = 0.4628, Log Rank

2. Secondary Outcome: Time to First Relapse During the Entire Double-Blind Treatment Period
Description: The time in days to first relapse is defined as the number of days from the date of randomization to the first relapse.
Time Frame: 104 Weeks
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Days
Groups:
- Rapastinel 450 mg Every 2 Weeks: Rapastinel 450 mg IV label once a week during OLTP followed by rapastinel 450 mg IV once every 2 weeks during DBTP.
Arm/Group | Placebo | Rapastinel 450 mg Every 2 Weeks | Rapastinel 450 mg Weekly
Number analyzed (Participants) | 202 | 202 | 200
Days | 232 [167 to 492] | 225 [127 to 323] | 336 [157 to NA] — Not enough events to allow the estimation of the percentiles and the standard error for the confidence intervals.
Statistical Analysis 1: Comparison: Placebo vs Rapastinel 450 mg Every 2 Weeks; Test type: Superiority; p = 0.6153, Log Rank
Statistical Analysis 2: Comparison: Placebo vs Rapastinel 450 mg Weekly; Test type: Superiority; p = 0.4123, Log Rank

3. Primary Outcome: Number of Participants Experiencing Suicidal Ideation or Suicidal Behavior Based on Columbia-Suicide Severity Rating Scale (C-SSRS) Using 5-Point Scales
Description: On the C-SSRS, the 5 types of suicidal ideation are:
  Type 1: "Wish to be dead" Type 2: Non-specific active suicidal thoughts Type 3: "Active suicidal ideation with any methods (not plan) without intent to act" Type 4: "Active suicidal ideation with some intent to act, without specific plan" Type 5: "Active suicidal ideation with specific plan and intent"
Time Frame: 104 Weeks
Population: The Double-blind modified Intent-to-Treat Population consists of all patients in the Open-label Safety Population who were randomized to a treatment group during the DBTP of the study and received at least 1 dose of IP during the DBTP. 1 subject in the Biweekly Rapastinel group did not have any responses regarding the C-SSRS during the DBTP.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Rapastinel 450 mg Every 2 Weeks | Rapastinel 450 mg Weekly
Number analyzed (Participants) | 202 | 201 | 200
Participants
  Suicidal Ideation | 17 | 25 | 23
  Suicidal Behavior | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: The study consisted of an 8 to 16 week OLTP; followed by a randomized DBTP of up to 104 weeks; followed by a 2 week safety period.
Arm/Group | OLTP Rapastinel 450 mg Weekly + ADT | DBTP Placebo | DBTP Rapastinel 450 mg Every 2 Weeks | DBTP Rapastinel 450 mg Weekly
All-Cause Mortality (participants affected / at risk) | 0/1304 | 1/202 | 0/202 | 0/200
Serious Adverse Events (participants affected / at risk) | 26/1304 | 6/202 | 3/202 | 5/200
Other Adverse Events (participants affected / at risk) | 290/1304 | 62/202 | 72/202 | 66/200
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | OLTP Rapastinel 450 mg Weekly + ADT (N=1304) | DBTP Placebo (N=202) | DBTP Rapastinel 450 mg Every 2 Weeks (N=202) | DBTP Rapastinel 450 mg Weekly (N=200)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 2 | 0 | 0 | 0
Major depression (Psychiatric disorders) | 2 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 1 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 2 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Endometrial hyperplasia (Reproductive system and breast disorders) | 1/920 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Lung carcinoma cell type unspecified recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 1/920 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Procedural vomiting (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Substance abuse (Psychiatric disorders) | 1 | 0 | 0 | 0
Substance use disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0 | 0
Traumatic liver injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 1
Device dislocation (Product Issues) | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1
Renal tubular necrosis (Renal and urinary disorders) | 0 | 0 | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Suicidal behaviour (Psychiatric disorders) | 0 | 0 | 0 | 1
Suicide threat (Psychiatric disorders) | 0 | 0 | 0 | 1
Ureterolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1
Anastomotic ulcer (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Breast cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1/54 | 0/60 | 0/48
Abscess intestinal (Infections and infestations) | 0 | 1 | 0 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Altered state of consciousness (Nervous system disorders) | 0 | 1 | 0 | 0
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | OLTP Rapastinel 450 mg Weekly + ADT (N=1304) | DBTP Placebo (N=202) | DBTP Rapastinel 450 mg Every 2 Weeks (N=202) | DBTP Rapastinel 450 mg Weekly (N=200)
Nasopharyngitis (Infections and infestations) | 79 | 15 | 16 | 15
Upper respiratory tract infection (Infections and infestations) | 73 | 19 | 16 | 25
Headache (Nervous system disorders) | 96 | 11 | 14 | 10
Dysgeusia (Nervous system disorders) | 89 | 5 | 14 | 2
Nausea (Gastrointestinal disorders) | 49 | 5 | 11 | 6
Diarrhoea (Gastrointestinal disorders) | 41 | 5 | 11 | 5
Bronchitis (Infections and infestations) | 12 | 5 | 5 | 10
Sinusitis (Infections and infestations) | 38 | 11 | 8 | 6
Weight increased (Investigations) | 37 | 4 | 11 | 3
Insomnia (Psychiatric disorders) | 52 | 11 | 10 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2018-11-06): https://cdn.clinicaltrials.gov/large-docs/88/NCT02951988/Prot_000.pdf
  • Statistical Analysis Plan (2018-12-13): https://cdn.clinicaltrials.gov/large-docs/88/NCT02951988/SAP_001.pdf